CLINICAL TRIAL: NCT06655090
Title: Fibrotic Interstitial Lung Disease Early Recognition and Strategic Therapy Study in China
Status: Recruiting | Type: Observational
Sponsor: Dai Huaping (Other)
Collaborators: The First Affiliated Hospital of Guangzhou Medical University (Other); Nankai University (Other); Jilin University (Other); Shanghai Pulmonary Hospital, Shanghai, China (Other); Shanghai Chest Hospital (Other); Institute of Basic Medical Sciences CAMS (Unknown); Tongji Hospital (Other); National Institute for Occupational Health and Poison Control (Unknown); Infervision Medical Technology Company Limited (Unknown)
Responsible Party: Sponsor-Investigator, Dai Huaping, Department of Pulmonary and Critical Care Medicine, China-Japan Friendship Hospital
Organization: China-Japan Friendship Hospital (Other)
Other Study IDs: ChinaJapanFH006
Record Dates: First submitted 2022-06-28; First posted 2024-10-23 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-07

CONDITIONS: Interstitial Lung Disease (ILD)
MeSH Terms: conditions — Lung Diseases, Interstitial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This project aimed to: 1) construct a cohort of no less than 10000 cases of f-ILD (including pneumoconiosis ≥3000 cases) with continuous regular follow-up to reveal the clinical phenotypes closely related to the development, progression and prognosis of pulmonary fibrosis; 2) systematically evaluate the safety and effectiveness of frozen lung biopsy, surgical lung biopsy/thoracoscopic lung biopsy and other techniques, and to optimize the histological diagnosis method of f-ILD; 3) construct a set of artificial intelligence (AI) evaluation system for quantitative evaluation of pulmonary fibrosis and its severity, and develop application software; 4) excavate and verify important molecular targets for the formation of pulmonary fibrosis and identify biomarkers; 5) combined with clinical phenotype, imaging, pathology and biomarkers to establish f-ILD early recognition and progress model, intervention strategies, guidelines and consensus, and applicated nationwide.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed as ILD

Exclusion Criteria:

* Lack of chest CT
* Patients refused to participant

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients were selected during hospitalization from medical organization.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Clinical diagnostic protocol of ILD tissue biopsy | 3 years
  Report on the reliability and safety assessment of TBLC and SLB diagnostics.
Predict model | 3 years
  The contents were based on the f-ILD cohort, combined with clinical, imaging, pathological, lung function and biomarker analysis, and constructed a multidimensional model for the early recognition and progression of f-ILD.
Severity of fibrosis in HRCT assessed by AI system in patients with ILD | 3 years
  Explore the diversity of abnormal image performance in patients with f-ILD, and extract multidimensional information based on deep learning and other methods. Realize the intelligent quantitative analysis of the severity of fibrosis.
F-ILD cohort | 6 years
  The researchers used inclusion/exclusion criteria for screening, and collected the demographic information, clinical symptoms and signs, laboratory tests, treatment, survival and other conditions of the patients who agreed to participate in the program and signed the informed consent, and collected biological specimens.
Important molecular targets and biomarkers identified by multi-omics | 3 years
  Single cell map of lung tissue in the early stage of ILD, key molecular targets and biomarkers for the development and progression of pulmonary fibrosis.

CONTACTS AND LOCATIONS:
Overall Officials: Huaping Dai, M.D. Ph.D., Study Director — China-Japan Friendship Hospital
Locations (1):
- China-Japan Friendship Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Wang S, Zhang X, Xie B, Ren Y, Geng J, Luo S, He X, Jiang D, He J, Hu Y, Zhu L, Li J, Zhou G, Liu M, Zhao L, Dai H. Fibrotic Interstitial Lung Disease Early Recognition and Strategic Therapy Study in China (FIRST): protocol for a prospective, multicentre registry study. BMJ Open. 2025 Nov 5;15(11):e105980. doi: 10.1136/bmjopen-2025-105980. PMID 41198211